CLINICAL TRIAL: NCT03134911
Title: Non-Interventional, Cross-sectional Study to Describe Health-related Quality of Life Among Controlled and Uncontrolled Patients With Nonvalvular Atrial Fibrillation on Anticoagulants. RE-QUOL Study.
Brief Title: Health-related Quality of Life in Patients on Anticoagulants
Acronym: RE-QUOL
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0280
Record Dates: First submitted 2017-03-01; First posted 2017-05-01 (Actual); Results first posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anticoagulation controlled patients: Treated with DOAC or VKA
  Interventions: Drug: DOAC or VKA
- anticoagulation non controlled patients: Treated with VKA
  Interventions: Drug: VKA

INTERVENTIONS:
Drug: DOAC or VKA — 6 months - 2 years
  Groups: anticoagulation controlled patients
Drug: VKA — 6 months - 2 years
  Groups: anticoagulation non controlled patients

SUMMARY:
The present study has been designed to describe the health-related quality of life in patients with non valvular atrial fibrillation who have been prescribed a specific anticoagulant treatment for their non valvular atrial fibrilation at least 6 months prior to study initiation. It will be conducted in Departments of Internal Medicine from approximately 50 centers in Spain. It consists of an only visit that will coincide with one of those performed by the patients as part of routine follow-up of their disease. 500 patients seen in internal medicine are planned to be included in the study

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and provides written informed consent to participate in this study.
* The patient is at least 18 years of age
* The patient has a diagnosis of non-valvular atrial fibrillation
* The patient is on the same anticoagulant therapy (VKA or DOAC) during at least 6 months and maximum 2 years.
* If treated with VKA, availability of % Time in Therapeutic Range (TTR) in past analytical records or enough amount of International Normalized Ratio (INR) measures to calculate it.

Exclusion Criteria:

* Current participation in any clinical trial of a drug or device
* Contraindication to the use of DOAC or VKA as described in the Summary of Product Characteristics (SmPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed of non valvular atrial fibrillation and prescribed DOACs or VKA, who are seen in internal medicine from hospitals of 3 Autonomous Communities in Spain (Madrid, Comunidad Valenciana, Andalucía)
Sampling Method: Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Canals, +34607550925, Study Chair — mireia.canals@boehringer-ingelheim.com
Locations (39):
- Spain (39):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares (Madrid)
  - HospitalUniversitario Príncipe de Asturias, Alcalá de Henares (Madrid)
  - Hospita Universitario Fundación Alcorcón, Alcorcón (Madrid)
  - Hospital Público Virgen de los Lirios, Alcoy (Alicante)
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario San Juan de Alicante, Alicante
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Universitario Monteprincipe, Boadilla Del Monte (Madrid)
  - Hospital San Juan de Dios, Bormujos (Sevilla)
  - Hospital General Universitario de Castellón, Castellón de La Plana (Castellón)
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario de Elche, Elche (Alicante)
  - Hospital Universitario de Fuenlabrada, Fuenlabrada (Madrid)
  - Hospital Comarcal Francesc de Borja, Gandía (València)
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital De Llíria (depende del Arnau de Vilanova), Llíria (Valencia)
  - Hospital de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hopital Clinico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda (Madrid)
  - Hospital Costa del Sol, Marbella (Málaga)
  - Complejo Hospitalario de Especialidades Virgen de la Victoria, Málaga
  - Hospital Regional de Málaga (Carlos Haya), Málaga
  - Hospital Universitario Rey Juan Carlos, Móstoles (Madrid)
  - Hospital Universitario de Móstoles, Móstoles (Madrid)
  - Hospital Vega Baja, Orihuela (Alicante)
  - Hospital Virgen del Camino, Pamplona (Navarra)
  - Hospital General de Requena, Requena (Valencia)
  - Hospital de Sagunto, Sagunto (Valencia)
  - Hospital Universitario Infanta Sofia, San Sebastián de Los Reyes (Madrid)
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario de Torrevieja, Torrrevieja (Alicante)
  - Hospital Clínico Universitariio de Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario de La Plana, Villarreal (Castellón)
  - Hospital Lluis Alcanyis, Xàtiva (Valencia)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational, multicentre and cross-sectional study conducted in Departments of Internal Medicine from 47 sites in Spain. The patient received the same anticoagulant treatment for at least 6 months and no more than 2 years.
Pre-assignment Details: Data were obtained from a single visit that coincided with one of those performed by the patients as part of routine follow-up of their disease, without interfering with usual clinical practice of the investigator. 535 patients were enrolled and 34 excluded from analysis due to being screening failure and not meeting inclusion/ exclusion criteria.
Groups:
- Total Patients With Non-valvular Atrial Fibrillation: Patients with non-valvular atrial fibrillation (NVAF) receiving conventional vitamin K antagonist (VKA) treatment with uncontrolled anticoagulation status and VKA or direct oral anticoagulant (DOAC) treatment with controlled anticoagulation status were included. For both the groups treatment were given for at least 6 months and up to 2 years.
Period: Overall Study
Arm/Group | Total Patients With Non-valvular Atrial Fibrillation
Started | 535
Completed | 501
Not Completed | 34
Not completed — Screen failure | 31
Not completed — Not meeting inclusion/exclusion criteria | 3

BASELINE CHARACTERISTICS:
Population: All patients with non-valvular atrial fibrillation (NVAF), who received conventional vitamin K antagonist (VKA) with uncontrolled anticoagulation status and those with controlled anticoagulation status receiving VKA or direct oral anticoagulant (DOAC) treatment at least 6 months and up to 2 years were included.
Groups:
- Uncontrolled Group: Patients with non-valvular atrial fibrillation (NVAF) receiving conventional vitamin K antagonist (VKA) treatment for at least 6 months and up to 2 years with uncontrolled anticoagulation status were included in this group.
- Controlled Group: Patients with non-valvular atrial fibrillation (NVAF), who received conventional vitamin K antagonist (VKA) or direct oral anticoagulant (DOAC) treatment for at least 6 months and up to 2 years with controlled anticoagulation status, were included in this group.
- Total: Total of all reporting groups
Arm/Group | Uncontrolled Group | Controlled Group | Total
Number analyzed (Participants) | 171 | 330 | 501
Age, Continuous [Mean (Standard Deviation); unit: Years] | 80.4 (8.7) | 79.3 (8.8) | 79.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 152 | 247
  Male | 76 | 178 | 254
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was not reported for this trial.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 171 | 330 | 501
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life (QoL) (HRQoL) Scores in the Spanish Adaptation of the Sawicki Questionnaire
Description: Sawicki questionnaire includes 32 items grouped in 5 dimensions: 1) general treatment satisfaction, 2) self-efficacy, 3) strained social network, 4) daily hassles and 5) distress. Patients estimated the impact of each item on their self-perceived treatment-related QoL on a scale of 1 (total disagreement) to 6 (total agreement). Response options for each question were: 1=not at all, 2=very little, 3=a little, 4=somewhat, 5=a lot, 6=very much. High scores in general treatment satisfaction and self-efficacy dimensions indicate high perceived HRQoL. Low scores in the strained social network, daily hassles and distress dimensions indicate high perceived HRQoL. The summary score for each dimension was calculated by dividing the total score of the sum of the items that comprise each dimension into the number of items included in that dimension. For the general treatment satisfaction dimension, the scores of individual questions have to be inverted first to calculate the dimension score.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Controlled Group | Uncontrolled Group
Number analyzed (Participants) | 330 | 171
Unit on scale
  Treatment satisfaction: number analyzed (Participants) | 321 | 166
  Treatment satisfaction | 4.9 (1.0) | 3.6 (1.3)
  Self-efficacy: number analyzed (Participants) | 321 | 166
  Self-efficacy | 4.3 (1.0) | 3.6 (1.0)
  Distress: number analyzed (Participants) | 319 | 166
  Distress | 3.1 (0.9) | 3.9 (1.1)
  Daily hassles: number analyzed (Participants) | 313 | 158
  Daily hassles | 2.1 (0.8) | 3.0 (1.0)
  Strained social network: number analyzed (Participants) | 317 | 163
  Strained social network | 1.8 (0.9) | 2.6 (1.2)

2. Secondary Outcome: Demographic Data of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Age group, work status and life status of uncontrolled non-valvular atrial fibrillation (NVAF) patients is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: All patients with non-valvular atrial fibrillation (NVAF), who received conventional vitamin K antagonist (VKA) treatment at least 6 months and up to 2 years with uncontrolled anticoagulation status were included.
Measure: Number; unit: Participants
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Participants
  Work status - Employed | 3
  Work status - Housewife | 40
  Work status - Retired | 126
  Work status - Other | 2
  Life status - Single | 8
  Life status - Married | 79
  Life status - Widowed | 78
  Life status - Divorced | 6
  Age < 65 | 10
  Age 65 - 75 | 32
  Age ≥ 75 | 129

3. Secondary Outcome: Height of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Height of uncontrolled non-valvular atrial fibrillation (NVAF) patients is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: All patients with non-valvular atrial fibrillation (NVAF), who received conventional vitamin K antagonist (VKA) treatment at least 6 months and up to 2 years with uncontrolled anticoagulation status were included. The number of patients included in the analysis of this variable has been specified.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 142
Centimeter (cm) | 163.1 (8.8)

4. Secondary Outcome: Weight of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Weight of uncontrolled non-valvular atrial fibrillation (NVAF) patients is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 144
Kilogram (kg) | 76.5 (16.1)

5. Secondary Outcome: Body Mass Index (BMI) of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: BMI of uncontrolled non-valvular atrial fibrillation (NVAF) patients is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram/meter^2 (kg/m^2)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 142
Kilogram/meter^2 (kg/m^2) | 28.7 (5.4)

6. Secondary Outcome: Kidney Function (Creatinine Clearance) of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Kidney function of uncontrolled non-valvular atrial fibrillation (NVAF) patients measured by creatinine clearance is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millilitre/minute (ml/min)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 150
Millilitre/minute (ml/min) | 57.2 (26.6)

7. Secondary Outcome: History of Non-valvular Atrial Fibrillation (NVAF) - Time Since Diagnosis
Description: Analysis of data regarding the specific NVAF profile of uncontrolled patients indicated that the average (± SD) time since diagnosis (calculated as the time from the date of diagnosis to the date of the baseline visit).
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Years | 2.5 (3.2)

8. Secondary Outcome: History of Non-valvular Atrial Fibrillation (NVAF) - Age at Diagnosis
Description: Age at diagnosis of uncontrolled non-valvular atrial fibrillation (NVAF) patients is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Years | 77.3 (8.7)

9. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Left ventricular ejection fraction (LVEF) of uncontrolled non-valvular atrial fibrillation (NVAF) patients is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 108
Percentage (%) | 56.1 (11.2)

10. Secondary Outcome: Percentage of Patients With Left Ventricular Ejection Fraction (LVEF) Depression of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Percentage of patients with left ventricular ejection fraction (LVEF) depression (% of LVEF depression) of uncontrolled non-valvular atrial fibrillation (NVAF) patients is presented qualitatively.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 161
Percentage of patients (%)
  Normal (≥ 50%) | 87.0
  Slightly depressed (41-49%) | 3.1
  Moderately depressed (31-40%) | 6.2
  Severely depressed (≤ 30%) | 3.7

11. Secondary Outcome: CHA2DS2-VASc Score of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: CHA2DS2-VASc stroke risk score is calculated based on the following conditions: Congestive heart failure, Hypertension, Age (≥ 75), Diabetes Mellitus, Stroke/ Transient Ischaemic Attack (TIA), Vascular disease, Age 65-74, Sex category. CHA2DS2-VASc stroke risk score may range from 0 to 9 with 0 being the best outcome.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Unit on scale | 4.5 (1.4)

12. Secondary Outcome: HAS-BLED Score of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: HAS-BLED bleeding risk score is calculated based on the following conditions: Hypertension, Abnormal renal and liver function, Stroke, Bleeding history or predisposition, Labile International Normalized Ratio (INR), Elderly (>65 years), Drugs and Alcohol. HAS-BLED bleeding risk score may range from 0 to 9 with 0 being the best outcome.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Unit on scale | 3.6 (1.1)

13. Secondary Outcome: Percentage of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients With History of Thromboembolic Events by Categories
Description: Percentage of uncontrolled non-valvular atrial fibrillation (NVAF) patients with history of thromboembolic events by categories are presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 60
Percentage of patients (%)
  Non-ST segment elevation myocardial infarction | 31.7
  Cerebral infarction | 28.3
  TIA | 21.7
  Pulmonary embolism | 8.3
  Stable angina pectoris | 6.7
  ST-segment elevation myocardial infarction | 6.7
  Unstable angina | 6.7
  Deep vein thrombosis | 5.0
  Systemic embolism | 1.7

14. Secondary Outcome: Percentage of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients With History of Haemorrhagic Events by Categories
Description: Percentage of uncontrolled non-valvular atrial fibrillation (NVAF) patients with history of haemorrhagic events by categories are presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 25
Percentage of patients (%)
  Gastrointestinal | 68.0
  Genitourinary | 12.0
  Pulmonary | 4.0
  Articular-muscular | 4.0
  Intracranial | 4.0
  Conjunctival | 4.0
  Nasal | 4.0

15. Secondary Outcome: Number of Visits to the Physician of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Number of visits to the internal medicine specialist per year of uncontrolled non-valvular atrial fibrillation (NVAF) patients is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Visits per year
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Visits per year | 3.1 (1.9)

16. Secondary Outcome: Therapeutic Time in Range (TTR%) of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Therapeutic time in range (TTR%) of uncontrolled non-valvular atrial fibrillation (NVAF) patients determined by the Rosendaal method (poor control < 65%) or by the direct method (poor control < 60%).
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Percentage (%)
  Rosendaal method (poor control < 65%): number analyzed (Participants) | 16
  Rosendaal method (poor control < 65%) | 49.1 (10.8)
  The direct method (poor control < 60%): number analyzed (Participants) | 155
  The direct method (poor control < 60%) | 35.0 (15.2)

17. Secondary Outcome: Time Since Treatment Initiation of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients
Description: Time since treatment initiation of uncontrolled non-valvular atrial fibrillation (NVAF) patients was calculated as the time from the start date of treatment to the date of the baseline visit.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Months | 14.8 (6.3)

18. Secondary Outcome: Percentage of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients Received Type of VKA Treatment
Description: Percentage of uncontrolled non-valvular atrial fibrillation (NVAF) patients received type VKA treatment is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Percentage of patients (%)
  Acenocoumarol | 97.7 (6.3)
  Warfarin | 2.3

19. Secondary Outcome: The Percentage of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients With Concomitant Diseases
Description: The percentage of uncontrolled non-valvular atrial fibrillation (NVAF) patients with at least one other concomitant diseases recorded in the medical history.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Percentage of patients (%)
  Hypertension: number analyzed (Participants) | 169
  Hypertension | 85.8
  Congestive heart failure: number analyzed (Participants) | 169
  Congestive heart failure | 48.5
  Diabetes mellitus: number analyzed (Participants) | 169
  Diabetes mellitus | 38.5
  Renal failure: number analyzed (Participants) | 169
  Renal failure | 34.3
  Anaemia: number analyzed (Participants) | 169
  Anaemia | 32.5
  Arterial vascular disease: number analyzed (Participants) | 169
  Arterial vascular disease | 19.5
  Previous stroke/transient ischaemic attack (TIA): number analyzed (Participants) | 169
  Previous stroke/transient ischaemic attack (TIA) | 17.8
  Venous thromboembolism: number analyzed (Participants) | 169
  Venous thromboembolism | 4.7
  Liver failure: number analyzed (Participants) | 169
  Liver failure | 1.8
  Other: number analyzed (Participants) | 169
  Other | 33.1

20. Secondary Outcome: The Percentage of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients With Active Concomitant Diseases on Visit Day
Description: The percentage of uncontrolled non-valvular atrial fibrillation (NVAF) patients with active concomitant diseases on visit day. The percentage was calculated on total patients who presented each of the diseases.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Percentage of patients (%)
  Hypertension | 72.5
  Congestive heart failure | 35.7
  Diabetes mellitus | 33.9
  Kidney failure | 28.1
  Anaemia | 25.1
  Arterial vascular disease | 10.5
  Previous stroke/TIA | 7.6
  Liver failure | 1.2
  Venous thromboembolism | 0.6
  Other | 23.4

21. Secondary Outcome: The Percentage of Uncontrolled Non-valvular Atrial Fibrillation (NVAF) Patients With Concomitant Treatment
Description: The percentage of uncontrolled non-valvular atrial fibrillation (NVAF) patients with concomitant treatment is presented.
Time Frame: The study consisted of a single visit between April 2017 and January 2018
Population: as for outcome 2
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Uncontrolled Group
Number analyzed (Participants) | 171
Percentage of patients (%)
  Yes | 97.1
  No | 2.9

ADVERSE EVENTS:
Time Frame: Adverse events collected during the study period between April 2017 and January 2018; up to 41 weeks
Groups:
- VKA Controlled Group: Patients with non-valvular atrial fibrillation (NVAF), who received conventional vitamin K antagonist (VKA) treatment for at least 6 months and up to 2 years with controlled anticoagulation status, were included in this group.
- DOAC Controlled Group: Patients with non-valvular atrial fibrillation (NVAF), who received direct oral anticoagulant (DOAC) treatment for at least 6 months and up to 2 years with controlled anticoagulation status, were included in this group.
Arm/Group | Uncontrolled Group | VKA Controlled Group | DOAC Controlled Group
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/69 | 0/261
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/69 | 1/261
Other Adverse Events (participants affected / at risk) | 0/171 | 0/69 | 0/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Uncontrolled Group (N=171) | VKA Controlled Group (N=69) | DOAC Controlled Group (N=261)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03134911/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT03134911/SAP_001.pdf